CLINICAL TRIAL: NCT03216772
Title: Safety and Efficacy of Using PK Morcellator With Pneumoliner Bag for Laparoscopic Morcellation With Laparoscopic Instrument for Tissue Containment and Removal During Laparoscopic Supracervical Hysterectomy or Total Laparoscopic Hysterectomy
Brief Title: Safety and Efficacy of Using PK Morcellator With Pneumoliner Containment Hysterectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was withdrawn for organizational reasons, not due to safety concerns.
Sponsor: Olympus Surgical Technologies Europe (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PK MORCELLATOR-LSH-01
Record Dates: First submitted 2017-07-08; First posted 2017-07-13 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Gynecologic Surgery
Keywords: Gynecologic Surgery; larscopy; morcellation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Olympus PK Morcellator in PneumoLiner (Experimental): Laparoscopic Supracervical Hysterectomy (LSH) or Total Laparoscopic Hysterectomy (TLH) using the Olympus PK Morcellator in PneumoLiner containment device
  Interventions: Device: Olympus PK Morcellator in PneumoLiner

INTERVENTIONS:
Device: Olympus PK Morcellator in PneumoLiner — Laparoscopic Supracervical Hysterectomy (LSH) or Total Laparoscopic Hysterectomy (TLH) using Olympus PK Morcellator in PneumoLiner containment device

SUMMARY:
The study is designed to evaluate the safety of performing in-bag morcellation of uterus tissues during laparoscopic hysterectomy (LSH or TLH). Pre- and perimenopausal women, aged 35-50 undergoing laparoscopic supracervical hysterectomy (LSH) or total laparoscopic hysterectomy (TLH)

ELIGIBILITY:
Inclusion Criteria:

* Pre- and Peri-menopausal woman patient age 35-50 years
* Women with fibroids and indication for laparoscopic hysterectomy at which a morcellators for cutting and extraction of tissue is required.
* Normal Pap test result in the last year
* Hemoglobin level of 10.0 g/dL or more at the time of treatment
* Subject able to comprehend and give informed consent for participation in this study
* Signed informed consent form

Exclusion Criteria:

* Patient is not considered suitable for a laparoscopic hysterectomy procedure
* Women with:
* Known or suspected gynecologic malignancy
* Known cervical dysplasia
* Postmenopausal women
* Undiagnosed vaginal bleeding
* Abdominal wall thickness is larger than 10 cm
* Atypical hyperplasia or malignancy in preoperative endometrial biopsy.
* Known cognitive disorder
* HIV or any other immunosuppressive disorder
* Liver disease
* Renal failure (Serum creatinine above 2.5 dL/ml)
* Cardiopulmonary disease contraindicating laparoscopic surgery
* History or evidence of gynecologic malignancy within the past five years
* Pace maker, internal defibrillator/cardio converter
* Impaired coagulation parameters
* Previous extensive pelvic surgery
* Psychological/psychiatric disease
* Contraindications to anesthesia or abdominal surgery.
* Concurrent participation in any other clinical study

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
The safety of using the PK MORCELLATOR in conjunction with the PneumoLiner containment device for contained cutting and extracting tissue during laparoscopic supracervical hysterectomy (LSH) or total laparoscopic hysterectomy (TLH). | End of study - approximately two years
  The safety of using the PK MORCELLATOR within the PneumoLiner containment bag for cutting and extracting tissue during LSH or TLH procedure will be determined by the probability of failure during in-bag morcellation procedure.
  * Failure is defined as "disruption of the isolation bag (using dye leak testing) or visible tissue dissemination".
  * Patient is defined "success" if no failure was detected as a result of the procedure.
  * Study safety success will be declared if no more than 1 failure (bag rapture) will be observed in 140 procedures.

SECONDARY OUTCOMES:
The efficacy of using PK MORCELLATOR in conjunction with the PneumoLiner containment device | End of study - approximately two years
  Ease of use of the PK MORCELLATOR in conjunction with the PneumoLiner containment device for LSH or TLH. Ease of use will be measured by designated Satisfaction Questionnaire.
Intra- or post-operative complications | End of study - approximately two years
  Intra or post complications rate (e.g. urinary, intestinal or nerve injury)
Mean procedure time | End of study - approximately two years
  Mean procedure time will be measured by hour/minutes.
Estimated blood loss during operation | End of study - approximately two years
  Blood loss during operation will be measured by volume (mL)
Post-operative pain | End of study - approximately two years
  Post-operative pain will be measured by Visual Analog Score - VAS
Hospitalization length | End of study - approximately two years
  Hospitalization length will be measured by days
Specimen weight | End of study - approximately two years
  Specimen will be measured by weight (gr)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Carey, MD, Principal Investigator — University of North Carolina, Chapel Hill

IPD SHARING:
Plan to Share IPD: No